CLINICAL TRIAL: NCT06600906
Title: Translating Hyperpolarized 13C MRI as a Novel Tool to Predict Treatment Response in Pancreatic Cancer
Brief Title: Hyperpolarized 13C MRI to Predict Response in Pancreatic Cancer
Status: Recruiting | Type: Observational
Sponsor: University of California, San Francisco (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Zhen Wang, MD, Principal Investigator, University of California, San Francisco
Other Study IDs: 24928; NCI-2024-07399 (Registry Identifier: NCI Clinical Trials Reporting Program (CTRP)); R01CA280071 (NIH)
Record Dates: First submitted 2024-09-14; First posted 2024-09-19 (Actual); Last update posted 2025-11-12 (Actual); Status verified 2025-11

CONDITIONS: Pancreatic Ductal Adenocarcinoma; Metastatic Pancreatic Ductal Adenocarcinoma; Locally Advanced Pancreatic Ductal Adenocarcinoma
MeSH Terms: interventions — Magnetic Resonance Spectroscopy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cohort A (HP 13C pyruvate, MRI): Participants with advanced/non-resectable pancreatic ductal adenocarcinoma (PDA) receive HP 13C pyruvate intravenously (IV) and undergo MRI scans prior to receiving standard-of-care (SOC) treatment and again at 4 weeks after starting SOC treatment. Participants may optionally undergo an additional HP 13C pyruvate MRI scan at 8 weeks after starting SOC treatment. Participants who have excellent response and deemed candidates for surgical resection may be switched to Cohort B. Participants also undergo CT and additional MRI scans throughout the study.
  Interventions: Drug: Hyperpolarized 13C-Pyruvate; Procedure: Computed tomography (CT); Procedure: Magnetic Resonance Imaging (MRI)
- Cohort B (HP 13C pyruvate, MRI): Participants with localized PDA who are deemed candidates for neoadjuvant therapy (NAT) receive HP 13C pyruvate IV and undergo MRI scans prior to starting NAT and again at 4 weeks after starting NAT. Participants may optionally undergo an additional HP 13C pyruvate MRI scan at 8 weeks after starting NAT. Participants who develop rapidly progressive disease and are deemed non-resectable may be switched to Cohort A. Participants also undergo CT and additional MRI scans throughout the study.
  Interventions: Drug: Hyperpolarized 13C-Pyruvate; Procedure: Computed tomography (CT); Procedure: Magnetic Resonance Imaging (MRI)

INTERVENTIONS:
Drug: Hyperpolarized 13C-Pyruvate — Given intravenously (IV)
  Other Names: HP 13C
Procedure: Computed tomography (CT) — Undergo CT imaging
  Other Names: CT
Procedure: Magnetic Resonance Imaging (MRI) — Undergo MRI imaging
  Other Names: MRI

SUMMARY:
This study evaluates an investigational scan called hyperpolarized carbon-13 pyruvate magnetic resonance imaging (MRI) in assessing treatment response in patients with pancreatic ductal carcinoma (PDA) that has spread to nearby tissue or lymph nodes (locally advanced) or that has spread from where it first started (primary site) to other places in the body (metastatic). MRI is a standard scan that helps doctors see tumors, organs, tissue, and bone. Standard contrast agents (e.g., gadolinium) are sometimes used to help make the scan images brighter, or easier to see. Hyperpolarized carbon-13 pyruvate is an experimental contrast agent that is different from standard MRI contrast in that it provides information on how a tumor processes nutrients. Hyperpolarized carbon-13 pyruvate MRI scans may work better than MRI with standard contrast agents in predicting how PDA tumors respond to treatment.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the percent changes in target tumor (primary tumor and/or abdominal metastases) hyperpolarized carbon C 13 pyruvate (HP 13C pyruvate) metabolism measures between the pre-treatment scan and the scan obtained 4 weeks (± 2 weeks) following treatment initiation. (Cohorts A and B).

II. To determine whether the changes in these metabolism measures are associated with best objective response (as defined by Response Evaluation Criteria in Solid Tumors [RECIST] version [v]1.1) on subsequent clinical computed tomography (CT) scans. (Cohorts A and B).

SECONDARY OBJECTIVES:

I. In patients who proceed to surgery following neoadjuvant therapy (NAT), to determine whether the HP 13C pyruvate metabolism in the primary tumor on the pre-operative MRI or the change in HP 13C pyruvate metabolism are associated with pathological response. (Cohort B).

II. To examine models from the primary objective where multiple imputation is used for where only pre-treatment imaging is available. (Cohorts A and B).

EXPLORATORY OBJECTIVES:

I. To determine whether the changes in target tumor (primary tumor and/or abdominal metastases) HP 13C pyruvate metabolism measures at 8 weeks (± 2 weeks) following treatment initiation are associated with best objective response as defined by RECIST v1.1 on subsequent clinical CT scans and clinical variables. (Cohort A).

II. To determine the repeatability of HP 13C pyruvate metabolism measures in the target tumor (primary tumor and/or abdominal metastasis) in patients with same-day repeated dose. (Cohorts A and B).

III. To compare the changes in HP 13C pyruvate metabolism measures to changes in tumor size and tumor apparent diffusion coefficients on the concurrently acquired 1H MRI. (Cohorts A and B).

IV. To determine whether the changes in target tumor (primary tumor and/or abdominal metastases) HP 13C pyruvate metabolism measures at 4 weeks (± 2 weeks) following treatment initiation (Cohorts A and B), 8 weeks (± 2 weeks) following treatment initiation (Cohort A), and after completion of NAT (Cohort B) are associated with progression-free survival (PFS) and overall survival (OS). (Cohorts A and B).

OUTLINE: Patients are assigned to 1 of 2 cohorts.

COHORT A: Patients with advanced/non-resectable pancreatic ductal carcinoma (PDA) receive HP 13C pyruvate intravenously (IV) and undergo MRI scans prior to receiving standard of care (SOC) treatment and again at 4 weeks after starting SOC treatment. Patients may optionally undergo an additional HP 13C pyruvate MRI scan at 8 weeks after starting SOC treatment. Patients who have excellent response and deemed candidates for surgical resection may be switched to Cohort B.

COHORT B: Patients with localized PDA who are deemed candidates for NAT receive HP 13C pyruvate IV and undergo MRI scans prior to starting NAT and again at 4 weeks after starting NAT. Patients may optionally undergo an additional HP 13C pyruvate MRI scan at 8 weeks after starting NAT. Patients who develop rapidly progressive disease and are deemed non-resectable may be switched to Cohort A.

Patients in both cohorts also undergo CT and additional MRI scans throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Participants must be 18 years or older.
* Histological or cytological confirmation of pancreatic ductal adenocarcinoma (PDA).
* Locally advanced or metastatic disease.
* At least one target lesion in the abdomen measuring ≥ 1centimeter (cm), according to RECIST v1.1.
* Eastern Cooperative Oncology Group (ECOG) Performance Status of 0, 1 or 2 (Karnofsky ≥ 50%)
* Participants with a prior or concurrent malignancy whose natural history or treatment does not have the potential to interfere with the safety or endpoints of this study are eligible.
* Ability to understand and willingness to sign a written informed consent document.

Exclusion Criteria:

* Participants unwilling or unable to undergo magnetic resonance (MR) imaging, including patients with contra-indications to MRI, such as cardiac pacemakers or non-compatible intracranial vascular clips.
* Poorly controlled hypertension, defined as either systolic > 170 or diastolic > 110. The addition of anti-hypertensives to control blood pressure is allowed for eligibility determination.
* Congestive Heart Failure ≥ Class III.
* Participants who are pregnant.
* Individuals of childbearing potential must agree to undergo a urine pregnancy test prior to participating in the study scans. Pregnant individuals are excluded because there is an unknown but potential risk for adverse effects in the unborn child secondary to administration of HP 13C pyruvate to the study participant. A female is considered to not be of childbearing potential (regardless of sexual orientation, having undergone a tubal ligation, or remaining celibate by choice), if they meet either of the following two criteria: (1) has reached a postmenopausal state (>= 12 continuous months of amenorrhea with no identified cause other than menopause); or (2) has undergone surgical sterilization (i.e., hysterectomy and/or bilateral oophorectomy for removal of uterus and/or ovaries).
* Participants who are breastfeeding/chestfeeding. Breastfeeding/chestfeeding individuals are excluded because there is an unknown but potential risk for adverse effects in the unborn/nursing child secondary to administration of HP 13C pyruvate to the study participant. Breastfeeding/chestfeeding should be discontinued before administration of HP 13C pyruvate.
* Known hypersensitivity to HP 13C pyruvate or any of its excipients.
* Participants with any condition or social circumstance that, in the opinion of the investigator, would impair the participant's ability to comply with study procedures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults receiving standard of care at University of California, San Francisco with biopsy-proven locally advanced or metastatic pancreatic ductal adenocarcinoma.
Sampling Method: Non-Probability Sample
Enrollment: 70 (Estimated)
Dates: Start 2024-10-01 (Actual); Primary Completion 2030-08-01 (Estimated); Study Completion 2032-09-01 (Estimated)

PRIMARY OUTCOMES:
Proportion of participants with best objective response (Cohorts A and B) | Up to 24 months
  The best objective response based on clinical imaging according to Response Evaluation Criteria in Solid Tumors (RECIST) version 1.11 will be reported
Mean percent change in target tumor peak HP 13C lactate/pyruvate ratio over time | Up to 6 weeks
  The mean percent change in peak HP 13C lactate/pyruvate ratio with 95% confidence intervals (CI) will be reported for scans completed at baseline and after 4 weeks (+/- 2 weeks) of non-interventional, standard of care treatment.
Mean change in target tumor HP 13C lactate/pyruvate area under the curve (AUC) ratio over time | Up to 6 weeks
  The mean change in HP 13C lactate/pyruvate area under the curve (AUC) ratio will be reported for scans completed at baseline and scans after 4 weeks (+/- 2 weeks) of non-interventional, standard of care treatment.
Mean percent change in target tumor HP 13C pyruvate to lactate conversion rate (kPL). | Up to 6 weeks
  The mean percent change in pyruvate to lactate conversion rate (kPL) will be reported for scans completed at baseline and scans after 4 weeks (+/- 2 weeks) of non-interventional, standard of care treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Zhen Wang, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No